CLINICAL TRIAL: NCT04953234
Title: A Pilot, Open-Label Study of NovoTTF-100L (TTFields, 150Hz) in Hospitalized Patients With COVID-19 and Continued Treatment After Hospitalization
Brief Title: Effect of Tumor Treating Fields (TTFields, 150 kHz) Concomitant With Best Standard of Care for the Treatment of Hospitalized COVID-19 Patients and Continued Treatment Following Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-37
Record Dates: First submitted 2021-07-04; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NovoTTF-100L (Experimental): Patients receive TTFields using the NovoTTF-100L System together with COVID-19 best standard of care
  Interventions: Device: NovoTTF-100L

INTERVENTIONS:
Device: NovoTTF-100L — Patients receive continuous TTFields treatment using the NovoTTF-100L device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the thorax. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields

SUMMARY:
The study is a prospective, pilot study aimed to test the safety of Tumor Treating Fields (TTFields) concomitant with best standard of care, for the treatment of hospitalized COVID-19 patients and continued treatment after hospitalization. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields) to the region of the organ to be treated, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

Tumor Treating Fields (TTFields) are a non-invasive, regional antimitotic treatment modality with minimal toxicity which have been approved for the treatment of recurrent and newly diagnosed glioblastoma (GBM) by the Food and Drug Administration (FDA) in the United States and have obtained a CE mark in Europe for the same indications. TTFields concomitant with chemotherapy were also approved for malignant pleural mesothelioma under FDA's humanitarian device exemption.

Cell culture study demonstrated that TTFields can significantly reduce corona virus infection and replication in human lung cells.

DESCRIPTION OF THE STUDY:

All patients included in this study are patients who are hospitalized due to COVID-19 disease. In addition, all patients must meet all eligibility criteria.

Eligible patients will be enrolled to the study and will receive COVID-19 best standard of care treatment concomitant with TTFields using the NovoTTF-100L System. The patients will be treated continuously with the device until discharge from the hospital and until there are no limitations on activities.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), attenuate SARS-CoV-2 virus infection and replication. TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTFields hold the promise of serving as a brand new treatment for COVID-19 disease with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Hospitalized with diagnosis of COVID-19 infection per reverse transcription polymerase chain reaction (RT-PCR) within 72 hours prior to treatment start.
3. SpO2 ≤ 93% at sea level.
4. Lung involvement confirmed with chest imaging.
5. Able and willing to comply with all study procedures.
6. Female participants of childbearing age must use highly effective contraception.
7. All patients must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

1. Receipt of any experimental treatment for COVID-19 prior to or during the study.
2. Assisted ventilation.
3. Critical illness: respiratory failure defined as oxygen saturation by pulse oximetry/inspired oxygen fraction (SpO2/FiO2) ratio < 150, septic shock, and/or multiple organ dysfunction.
4. Significant co-morbidities at baseline as determined by the investigator:

   1. Clinically significant hematological, hepatic and renal dysfunction, defined as: Neutrophil count < 1.5 x 10^9/L and platelet count < 100 x 10^9/L; bilirubin > 1.5 x upper limit of normal (ULN); aspartate aminotransferase (AST) and/or alanine transaminase (ALT) > 2.5 x ULN; and serum creatinine > 2.5 mg/dL.
   2. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class IV (unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases).
   3. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the study.
   4. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent.
5. Implantable electronic medical devices (e.g. pacemaker, defibrillator) in the upper torso.
6. Pregnancy or breast-feeding.
7. Known allergies to medical adhesives or hydrogel.
8. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's cooperation or other unspecified reasons that, in the opinion of the Investigator or sponsor, make the subject's enrollment incompatible with study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | 2 months

SECONDARY OUTCOMES:
All-cause mortality | Day 1 through Day 29
  The proportion of participants who died by study Day 29.
Incidence of intensive care unit admission | Day 1 through Day 29
Incidence of non-invasive ventilation or high-flow oxygen use | Day 1 through Day 29
Incidence of invasive ventilation | Day 1 through Day 29
Incidence of extracorporeal membrane oxygenation | Day 1 through Day 29
Patient inflammatory status | Day 3, 8, and 11
  Inflammatory status measured as the difference in C reactive protein (CRP), D-dimer and ferritin blood levels from baseline on days 3, 8 and 11 until discharge.
Duration of hospitalization | Day 1 through Day 29
Time to recovery | Day 1 through Day 29
  Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale: 1) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Not hospitalized, no limitations on activities.
Clinical status at day 8, 15, 22, 29 | Day 8, 15, 22, and 29
  Clinical status according to ordinal scale. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided